CLINICAL TRIAL: NCT06128265
Title: Sleep Extension or Regularity to Reduce Diabetes Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1060
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, randomized and unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Extension (Experimental): Participants that are in the sleep extension group will have their time in bed extended by 2 hours. This can include going to bed earlier and/or waking up later.
  Interventions: Behavioral: Sleep Extension
- Sleep Regularity (Experimental): Participants in the sleep regularity group will have consistent bedtimes (within 30min).
  Interventions: Behavioral: Sleep Regularity

INTERVENTIONS:
Behavioral: Sleep Extension — Extending time in bed by 2 hours (going to bed earlier and/or waking up later)
  Arms: Sleep Extension
Behavioral: Sleep Regularity — Consistent bedtimes (within 30min)
  Arms: Sleep Regularity

SUMMARY:
The goal of this study is to identify an intervention that improves sleep health and consequently metabolic health by examining whether sleep extension or enforced regularity in short sleepers will have beneficial effects on diabetes and obesity risk.

DETAILED DESCRIPTION:
Numerous studies of restricted sleep have revealed insufficient sleep as a novel risk factor for metabolic disease. Specifically, it has been reported that insufficient sleep resulted in impairments in appetite regulation, energy intake, glucose tolerance, and insulin sensitivity. Further, recent studies have begun to reveal that the regularity of sleep timing may also impact metabolic health, in that increased sleep variability was associated with greater cardio-metabolic risk. Alternatively, only a few studies have explored whether sleep extension could be beneficial to metabolic outcomes, and no studies have focused on improved regularity or racial disparities. These studies have revealed improvements in glucose metabolism and caloric intake in predominantly non-Hispanic White individuals. Therefore, in this pilot study, we seek to examine whether sleep extension or enforced regularity can improve diabetes and obesity risk in a population known to be differentially impacted by sleep deficiency and metabolic disease, short sleeping African American and Black adults.

The investigator proposes to first assess sleep duration, food intake, ratings of hunger/appetite and reward-related eating, daily interstitial glucose, resting metabolic rate, insulin sensitivity, and glucose tolerance in short sleeping overweight African American and Black adults during a baseline/habitual sleep assessment. Participants will then be randomized to one of two different 14-day sleep interventions: sleep extension or sleep regularity. Following the intervention, assessments of food intake, ratings of hunger/appetite and reward-related eating, daily interstitial glucose, resting metabolic rate, insulin sensitivity, and glucose tolerance will be repeated. The goal of this pilot project is to demonstrate feasibility of our study design, particularly effectively impacting sleep in the home. The aims of this pilot study are to demonstrate:

1. that participants can extend sleep by ~2 hours or adhere to sleep regularly within a 30min window at home for two weeks,
2. changes in glucose metabolism following the interventions and
3. changes in subjective hunger/appetite ratings and food intake

This experimental approach is expected to reveal novel and important interventions that can have a beneficial impact on the risk of diabetes and obesity in an understudied population that suffers from increased risk, short sleeping overweight African American and Black adults.

ELIGIBILITY:
Inclusion Criteria:

* African American or Black men and women
* Age 21-50 years old
* Overweight (BMI greater than or equal 25 kg/m2 and less than 35 kg/m2)
* Self-reported short sleep (less than 7hrs/night, sleep between 22:00-08:00, and who indicate they could sleep more if they had the opportunity)
* No previously diagnosed sleep disorders (including obstructive sleep apnea (OSA))
* No existing diagnosis of diabetes
* No history of endocrine dysfunction
* No history of psychiatric, cardiovascular, or eating disorders, not having a gastro-intestinal disease that requires dietary adjustment,
* Currently taking no medications (excluding statins and birth control)

Exclusion Criteria:

* Drug and nicotine use
* Habitual alcohol use of more than 2 drinks per day
* Caffeine intake of more than 500 mg per day
* Subjects who participated in medically managed weight loss program within the past year
* Subjects who have undergone bariatric surgery,
* Subjects who have dietary restrictions,
* Subjects who worked night shifts, or crossed any time zones in the month prior to the study.
* Sleep-disordered breathing (apnea-hypopnea index>15 events/hour) from an overnight at home sleep test (NOX)
* Peri- and post-menopausal women will not be included.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep outcome measures- Sleep time | Baseline to Day 24
  A decrease in time to sleep onset from baseline to day 24 measured in time of day by Wrist Actigraphy Monitoring.
Sleep Outcome- Wake time | Baseline to Day 24
  Change in wake time from baseline to day 24 measured in time of day by Wrist Actigraphy Monitoring.
Sleep outcome- Sleep duration | Baseline to Day 24
  Change in Sleep duration from baseline to day 24 measured in minutes by Wrist Actigraphy Monitoring.
Sleep Outcome- Regularity of sleep | Baseline to Day 24
  Change in regularity of sleep from baseline to day 24 measured by Wrist Actigraphy Monitoring. The value is from standard deviation of time of middle of the sleep period.
Sleep Outcome- Sleep Efficiency | Baseline to Day 24
  Change in sleep efficiency from baseline to day 24 measure by a percentage of total sleep time/time in bed from Wrist Actigraphy Monitoring.
Change in glucose homeostasis after 24 days | Baseline to Day 24
  The Matsuda Index of whole body insulin sensitivity, the homeostasis model assessment (HOMA) measures beta cell function and insulin resistance will be measured by Oral glucose tolerance test (OGTT).
Change in glucose homeostasis measured by Continuous Glucose Monitor (CGM) | Baseline to Day 24
  Mean Absolute Glucose (MAG - mg/dl), Coefficient of Variation (CV - mg/dl), Standard Deviation (SD-mg/dl), Area Under the Curve (AUC - mg/dl), Time Spent in Range (TIR - minutes), Continuous Overall Net Glycemic Action (CONGA - (mg/dl) per minutes) will be measured by Continuous Glucose Monitor (CGM).

SECONDARY OUTCOMES:
Changes from baseline through day 24 of novel Patient Reported Outcome instrument | Baseline to Day 24
  Detection of within-patient changes in sleep effects (sleepiness), appetite, mood, reported in a novel Patient-Reported Outcome instrument between baseline and Day 24.
Glucose Homeostasis-First phase insulin response | Baseline to Day 24
  Changes in first phase insulin response (ARIg=mu.i^-1.min) from baseline to Day 24 measured by oral glucose tolerance test (OGTT).
Glucose Homeostasis-Oral disposition index (DIo) | Baseline to Day 24
  Changes in oral disposition index (DIo) from baseline to Day 24 measured in (SI x ARIg = [(mu/l)^-1.min^-1] * [mu.l^-1.min]) by oral glucose tolerance test (OGTT).
Glucose Homeostasis- insulinogenic index | Baseline to Day 24
  Changes in insulinogenic index (change in plasma insulin/change in plasma glucose from 0-30 minutes = (pmol/L)/(mg/dL)) from baseline to Day 24 measured by oral glucose tolerance test (OGTT).
Weight in kg, measured from screening through study completion. | Screening to Day 24
  The change in weight values will be measured by in laboratory anthropometrics measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hanlon, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
A limited data set will be shared with a collaborator at the University of Northwestern.